CLINICAL TRIAL: NCT03135886
Title: A Cluster RCT to Increase HIV Testing in Substance Use Treatment Programs
Brief Title: Project I Test: Implementing HIV Testing in Opioid Treatment Programs
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Weill Medical College of Cornell University (Other); University of Miami (Other); Boston Medical Center (Other); Research Foundation for Mental Hygiene, Inc. (Other); San Francisco Department of Public Health (Other Government); New York University Abu Dhabi (Other)
Responsible Party: Principal Investigator, Lisa Metsch, Professor of Sociomedical Sciences, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAQ9986; R01DA043130 (NIH)
Record Dates: First submitted 2017-04-26; First posted 2017-05-02 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: HIV/AIDS; Hepatitis C; Substance Use Disorders; Opioid-use Disorder
Keywords: HIV; HIV Testing; Hepatitis C Virus Testing; Opioid Use Disorder Treatment; Substance Use Disorders Treatment; Hepatitis C Virus; Practice Coaching
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C; Substance-Related Disorders; Opioid-Related Disorders | interventions — Seroconversion

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized controlled trial (RCT) where approximately 51 sites will be randomly inducted into the study. Site randomization to condition will occur on a rolling basis in intervals of approximately 14-18 days. Selected sites will be invited to participate in the study and randomly assigned to one of the three conditions (described below).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HIV Testing Practice Coaching Intervention Group (Experimental): The HIV Testing Practice Coaching (PC) Intervention is designed to improve the provision and sustained implementation of on-site HIV testing and linkage to care among OTP patients.
  Interventions: Other: HIV Testing Practice Coaching Intervention
- HIV and HCV Testing Practice Coaching Intervention Group (Experimental): The HIV and HCV Testing Practice Coaching (PC) Intervention will leverage the HIV PC intervention and follow the same interventional steps described above, and, in addition, provide information and training to support joint HIV/HCV testing and linkage to care among OTP patients.
  Interventions: Other: HIV and HCV Testing Practice Coaching Intervention
- Information Control Group (Other): The administrators of OTPs assigned to the control condition will receive a website link to and hard copy of the NIDA/SAMHSA Blending Initiative product for HIV rapid testing.
  Interventions: Other: Information Control

INTERVENTIONS:
Other: Information Control — The OTPs assigned to this group will be provided access to the NIDA/SAMHSA Blending Initiative product for HIV rapid testing. Resources generated from the HIV rapid testing Blending Initiative product include a fact sheet, resource guide, marketing materials, and an Excel-based budgeting tool. In addition to the HIV-specific materials, the website provides opportunities for training, self-study progress, workshop, and distance learning. OTPs also will receive a link to the Anti-Retroviral Treatment and Access to Services (ARTAS) intervention training website which provides information and training courses. Sites also will receive a hard (or electronic) copy of the ARTAS implementation manual and information about the provision of HIV testing, linkage to care and PrEP.
  Arms: Information Control Group
Other: HIV and HCV Testing Practice Coaching Intervention — The practice coaches (PCs) will work with the program team a) to establish capabilities, reimbursement systems and/or partnerships necessary to support HIV and HCV testing and evidence--based linkage to care and b) to reduce barriers (e.g., staffing, training) to the implementation and sustained provision of HIV and HCV testing. Also, due to the expense of HCV treatment, and potentially more complicated mechanisms for linking HCV-positive patients to further evaluation and care which may take more time than anticipated, PCs will provide OTPs with basic education and motivation about the importance of HCV testing for reasons other than immediate curative treatment. Information on PrEP also will be provided. The intervention will occur over approximately 29 weeks (or 6 months).
  Arms: HIV and HCV Testing Practice Coaching Intervention Group
Other: HIV Testing Practice Coaching Intervention — The practice coaches (PCs) will work with the programs a) to establish capabilities, reimbursement systems and/or partnerships necessary to support HIV testing and evidence-based linkage to care and b) to reduce barriers (e.g., staffing, training) to the implementation and sustained provision of HIV testing. Information on Pre-Exposure Prophylaxis (PrEP) also will be provided. The intervention will occur over approximately 29 weeks (or 6 months) consisting of four distinct evidence-based phases designed to establish competency in the implementation of organizational change towards establishing HIV testing outcomes among OTP clientele.
  Arms: HIV Testing Practice Coaching Intervention Group

SUMMARY:
This study will test two active evidence-based "practice coaching" (PC) interventions to improve opioid treatment programs' (OTPs') provision and sustained implementation of on-site 1) HIV testing and linkage to care and 2) HIV/Hepatitis C virus (HCV) testing and linkage to care among patients seeking/receiving substance use disorder treatment.

Aims are:

Aim 1: To evaluate the effectiveness of the PC interventions on improving patient uptake of HIV testing in OTPs including the incremental impact of the HIV/HCV intervention on HIV testing.

Aim 2: To examine, using mixed-methods, the impact of the PC interventions on the initiation and sustained provision of HIV testing and timely linkage to care.

Aim 3: To evaluate the health outcomes, health care utilization, and cost-effectiveness of the PC interventions compared incrementally to one another and to the control condition.

Primary Hypothesis:

1. The two PC interventions will result in significantly higher proportions of patients tested for HIV than the information control condition during the "initial impact" period (7-12 months post-randomization or T3), controlling for the proportion of patients tested during the baseline period, T1 (Primary) and during the "sustained impact" period, 13-18 months post-randomization or T4 (Secondary).
2. The HIV/HCV PC intervention will result in significantly higher proportions of patients tested for HIV than the HIV PC intervention during the initial impact period (7-12 months post-randomization or T3), controlling for the proportion of patients tested during the baseline period, T1 (Secondary) and during the "sustained impact" period, 13-18 months post-randomization or T4 (Secondary).

DETAILED DESCRIPTION:
Using the most recent National Survey of Substance Abuse Treatment Services (N-SSATS) data available from the Substance Abuse and Mental Health Services Administration (SAMHSA) as the sampling frame, 51 sites will be randomly selected to participate in the study. Site randomization to condition will occur on a rolling basis. Selected sites will be invited to participate in the study and randomly assigned to one of the three intervention conditions (17 sites per condition) -- information control, HIV PC, and HIV/HCV PC. The control condition will be an HIV testing informational product consisting of the official NIDA/SAMHSA Blending Initiative product, "HIV Rapid Testing in Substance Abuse Treatment Programs," ARTAS intervention information and Pre-Exposure Prophylaxis (PrEP) information that will be provided to OTPs to educate and motivate them about the importance of offering on-site HIV testing and linkage to care. In the active PC conditions, champions and key OTP staff will be provided coaching and support for the implementation of an innovation (i.e., offering HIV testing on-site and linking persons living with HIV to care) and for sustaining resulting improvements in testing.

De-identified aggregate client data on HIV and HCV testing and linkage to care will be provided by the sites for four 6-month-long time intervals: T1 (up to 6 months prior to randomization), T2 (during the intervention/control period, up to 6 months post-randomziation), T3 (7-12 months post-randomization), and T4 (13-18 months post-randomization). Qualitative and quantitative site-level data will also be collected immediately preceding randomization and again during interval T3.

ELIGIBILITY:
Inclusion Criteria:

* Eligible sites must:

  1. See at least 150 unduplicated patients/year/site
  2. Be capable and willing to prospectively collect data on the number of patients who a) are offered any HIV and/or HCV tests; b) completed these tests; c) are referred to care/evaluation (and type of referral) if positive; and d) are linked to care/evaluation within 30 days of diagnosis
  3. Be capable and willing to provide patient demographics, testing data within demographic categories of gender and race/ethnicity (in aggregate) and data on HIV/HCV test reimbursement processes and outcomes
  4. Have key staff willing to consent to participate in study surveys, qualitative interviews and intervention coaching throughout the study

Exclusion Criteria:

* Sites will be excluded if:

  1. Over 50% of patients served in the prior 6 months were HIV or HCV tested
  2. They are terminated via PI decision/discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 418 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of OTP patients HIV tested at 6 months post intervention or control, while controlling for HIV testing during the baseline period (T1) | The period 7-12 months post site-randomization (T3).
  The primary outcome measure will be a contrast of the proportion of OTP patients HIV tested during T3, controlling for HIV testing at baseline (T1). The primary test will be whether the proportion of patients tested across the two PC interventions--HIV Testing PC Intervention Group and HIV/HCV Testing PC Intervention Group--differs from the proportion of patients tested in the Information Control Group.

SECONDARY OUTCOMES:
Proportion of OTP patients HIV tested at 12 months post intervention or control | The period 13-18 months post site-randomization.
  The secondary outcome measure will be the proportion of OTP patients HIV tested during T4, controlling for HIV testing at baseline (T1). One test will be whether the proportion of patients tested across the two PC interventions--HIV Testing PC Intervention Group and HIV/HCV Testing PC Intervention Group--differs from the proportion of patients tested in the Information Control Group. A second test will be whether the proportion of OTP patients HIV tested during T4 in the HIV Testing PC Intervention Group differs from the proportion of patients tested in the HIV/HCV Testing PC Intervention Group.

OTHER OUTCOMES:
OTPs' incremental cost-effectiveness ratio (ICER) | 6 months post randomization (T2).
  The ICER is a statistic used to summarize the cost-effectiveness of a health care intervention and is defined by the difference in cost between two possible interventions, divided by the difference in their effect. One ICER will be calculated for the difference between the Information Control Group and HIV Testing PC Intervention Group. A second ICER will be calculated for the difference between the HIV Testing PC Intervention Group and the HIV/HCV Testing PC Intervention Group.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Metsch, PhD, Principal Investigator — Columbia University; Daniel Feaster, PhD, Principal Investigator — University of Miami; Jemima Frimpong, PhD, Principal Investigator — New York University Abu Dhabi; Lauren Gooden, PhD, Study Director — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The data and associated documentation may become available to other researchers under a data-sharing agreement. All interested researchers must contact the PI and provide a proposal explaining the analysis that will be conducted and specify which IPD is needed to accomplish this.

REFERENCES:
- [Background] Frimpong JA, Parish C, Feaster DJ, Gooden LK, Matheson T, Haynes L, Linas BP, Assoumou SA, Tross S, Kyle T, Nelson CM, Liguori TK, Toussaint O, Siegel K, Annane D, Metsch LR. A study protocol for Project I-Test: a cluster randomized controlled trial of a practice coaching intervention to increase HIV testing in substance use treatment programs. Res Sq [Preprint]. 2023 Jun 28:rs.3.rs-3059783. doi: 10.21203/rs.3.rs-3059783/v1. PMID 37461594
- [Derived] Frimpong JA, Parish CL, Feaster DJ, Gooden LK, Nelson MC, Matheson T, Siegel K, Haynes L, Linas BP, Assoumou SA, Tross S, Kyle T, Liguori TK, Toussaint O, Annane D, Metsch LR. A study protocol for Project I-Test: a cluster randomized controlled trial of a practice coaching intervention to increase HIV testing in substance use treatment programs. Trials. 2023 Sep 26;24(1):609. doi: 10.1186/s13063-023-07602-8. PMID 37749635
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37461594/